CLINICAL TRIAL: NCT02620917
Title: Survey on Continuos Subcutaneous Insulin Infusion in Italy
Brief Title: Continuos Subcutaneous Insulin Infusion in Italy
Acronym: IMITA2
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Daniela Bruttomesso, MD medical doctor, PhD, University of Padova
Other Study IDs: 3506/AO/15
Record Dates: First submitted 2015-11-23; First posted 2015-12-03 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; CSII
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, multicenter, cross sectional study, collecting clinical and metabolic informations about patients treated with CSII in Italy.

DETAILED DESCRIPTION:
The aim of the study is to collect clinical and metabolic characteristics of patient treated with CSII in Italy.

Data will be collected through a questionnaire sent by e-mail to CSII experienced Diabetes Centers ( both adult and pediatric patients) . The questionnaire assessed: (1) number of CSII-treated patients; (2) patients and pump characteristics; (3) structure and organization of Diabetes Centers providing CSII therapy; (4) metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* all patients treated with CSIIin Italy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: we will evaluate allItalian patients treated with insulin pump
Sampling Method: Non-Probability Sample
Enrollment: 6623 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bruttomesso, MD, PhD, Principal Investigator — University of Padova
Locations (1):
- University of Padova, Padua, Italy

REFERENCES:
- [Derived] Lepore G, Bonfanti R, Bozzetto L, Di Blasi V, Girelli A, Grassi G, Iafusco D, Laviola L, Rabbone I, Schiaffini R, Bruttomesso D; Italian Study Group on the Diffusion of CSII. Metabolic control and complications in Italian people with diabetes treated with continuous subcutaneous insulin infusion. Nutr Metab Cardiovasc Dis. 2018 Apr;28(4):335-342. doi: 10.1016/j.numecd.2017.12.001. Epub 2017 Dec 9. PMID 29428572

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Subcutaneous Insulin Infusion (CSII) Treatment: Patients who received Continuous subcutaneous insulin infusion (CSII) treatment in Italy
Period: Overall Study
Arm/Group | Continuous Subcutaneous Insulin Infusion (CSII) Treatment
Started | 6623
Completed | 6623
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CSII Treatment: Patients who received CSII treatment in Italy
Arm/Group | CSII Treatment
Number analyzed (Participants) | 6623
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [22 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3827
  Male | 2796
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6623
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 6623

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Assessed by Median of HbA1c,
Description: median of HbA1c measured in the last year
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: mmol/mol
Arm/Group | CSII Treatment
Number analyzed (Participants) | 6623
mmol/mol | 60 [53 to 67]

2. Primary Outcome: Patients With Severe Hypoglycemia
Description: Number of patients reporting severe hypoglycemia (requiring assistance by an other person) in the last year
Time Frame: 1year
Measure: Number; unit: participants
Arm/Group | CSII Treatment
Number analyzed (Participants) | 6623
participants | 331

3. Primary Outcome: Number of Patients With Glycated Hemoglobin on Target
Description: number of patients who achieved HbA1c target (< 7,5% in patients < 18 years old; <7% in adult patients);
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Adults on CSII Treatment: Patients who received CSII treatment in Italy ( = or > 18 YEARS OLD)
- Paediatric Patients on CSII Treatment: Patients < 18 years old ON CSII treatment
Arm/Group | Adults on CSII Treatment | Paediatric Patients on CSII Treatment
Number analyzed (Participants) | 5598 | 1025
participants | 1288 | 445

4. Secondary Outcome: Number of Patients With HbA1c on Target Using Advanced Pump's Functions, CGM and CHO Counting
Description: number of patients adults with HbA1c <7,0% using advanced pump's functions, CGM and CHO counting number of paediatrics patients with HbA1c < 7.5% using advanced pump's functions, CGM and CHO counting
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Adults on CSII Treatment | Paediatric Patients on CSII Treatment
Number analyzed (Participants) | 5598 | 1025
participants | 1713 | 515

ADVERSE EVENTS:
Time Frame: time of observations= 1 years.
Description: no adverse events (study correlated and not study correlated) occurred
Arm/Group | CSII Treatment
All-Cause Mortality (participants affected / at risk) | 0/6223
Serious Adverse Events (participants affected / at risk) | 0/6223
Other Adverse Events (participants affected / at risk) | 0/6223

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02620917/Prot_SAP_000.pdf